CLINICAL TRIAL: NCT05601570
Title: Impact of the Experience of Anaesthetists in Changing Ventilation Strategies During Panendoscopy on the Incidence of Intraoperative Hypoxaemia
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, David Ferreira, Principal Investigator, Centre Hospitalier Universitaire de Besancon
Other Study IDs: ID020621HFNO
Record Dates: First submitted 2022-10-23; First posted 2022-11-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: ENT Tumor
Keywords: Panendoscopy; High Flow Nasal Oxygen; face mask ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
High Flow Nasal Oxygen Therapy (HFNO) is a new oxygenation tool that is becoming increasingly widespread in perioperative anaesthesia. The benefits of this oxygenation tool are based on different physiological principles. These include the reduction of dead space by "flushing" the nasopharyngeal cavities, positive airway pressure and the warming and humidification of inspired air. In addition, the high flow rates used ensure that the patient's inspiratory demand is covered, allowing for the delivery of oxygen-enriched and controlled air. It is simple to use, with the only parameters to be set being gas flow and FiO2. The use of HFNO appears to allow a prolongation of apnoea time without desaturation in apneic ventilation.

Mainly studied in ENT surgery because of the interest that this oxygenation strategy presents with the absence of recourse to oro-tracheal intubation (OTI), several authors will use it in the framework of micro-laryngoscopy surgery in suspension. However, its use as an oxygenation strategy during panendoscopy has been little explored. Panendoscopy is a common procedure that requires deep and short anesthesia. The main challenge is the sharing of the airway between the anesthesia team and the surgical team. Learning to use this new method or the impact of operator experience has never been explored.

DETAILED DESCRIPTION:
Currently, there are several strategies to ensure oxygenation during this specific type of ENT management:

* Mechanical ventilation with oro-tracheal intubation (OTI)
* Face mask ventilation (FMV)
* Jet ventilation
* HFNO Each of these methods has advantages and disadvantages, which explains why there are no clear recommendations to date on the preferred anesthesia and oxygenation technique. Regardless of the method chosen, the risks remain significant for the patient, particularly the risk of hypoxemia during a desaturation episode.

For several years, the strategy of oxygenation during panendoscopy and the number of practitioners performing this procedure has evolved in our centre.

* 2017, with the arrival of the HFNO in the operating room.
* 2020, during the SARS-CoV2 pandemic, changes in the organisation of the anaesthesiology department had to take place and the number of practitioners performing this procedure increased significantly.

The main objective of this study was to evaluate the impact of the evolution periods of the oxygenation strategies and the experience of the operators on the incidence of patients with at least one intra-procedural hypoxemia (SpO2 < 90% for more than one minute).

All patients who had a panendoscopy from 01 January 2015 to 31 December 2020 were analysed. The anaesthetists in our centre are divided into different practice specialties, so a small number of them regularly perform anaesthesia in ENT surgery. We divided the anaesthetists who performed panendoscopies during the study period into two categories in order to compare the incidence of severe hypoxaemia (SpO2 < 90%) among them :

* Experienced anaesthetists (practitioner who has performed at least 30 panendoscopies per year for two consecutive years)
* Non-experienced anaesthetists (practitioner who has performed at least one panendoscopy per year and does not meet the criteria for expertise)

ELIGIBILITY:
Inclusion Criteria:

* major patients receiving panendoscopy

Exclusion Criteria:

* panendoscopies performed in combination with another invasive procedure that may alter anaesthetic management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All major patients receiving panendoscopy during the period 2015 - 2020 in our center
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with oxygen desaturation | during the intervention (max 6hours)from induction of anaesthesia to discharge from the operating theatre
  Proportion of patients with oxygen desaturation (SpO2 < 90%) for more than 1 minute.

SECONDARY OUTCOMES:
Proportion of patients within each of the ventilation modalities used in panendoscopies | during the intervention (max 6hours)from induction of anaesthesia to discharge from the operating theatre
  Proportion of patients within each of the ventilation modalities used in panendoscopies Proportion of patients requiring repeat face mask ventilation (at least one reventilation outside the initial denitrogenation)
Proportion of patients requiring oro-tracheal intubation
  Proportion of patients intubated during panendoscopy
Duration of the procedure | during the intervention (max 6hours)from induction of anaesthesia to discharge from the operating theatre
  Time (minutes) from induction of anaesthesia to discharge from the operating room
Incidence of major intraoperative complications | during the intervention (max 6hours)from induction of anaesthesia to discharge from the operating theatre
  Complications are : Extreme bradycardia < 30 beats per minute, hemodynamic instability defined by MAP < 40 mmHg, hypercapnia (more than 80 mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, Franche Comté, France